CLINICAL TRIAL: NCT00521716
Title: A Single Arm, Uni-Center, Prospective Clinical Investigation to Evaluate Safety and Efficacy of the WaisFix100i for Intracapsular Femoral Fracture Fixation
Brief Title: Safety and Efficacy of the WaisFix100i for Intracapsular Femoral Fracture Fixation
Status: Suspended | Phase: Not Applicable | Type: Interventional
Sponsor: OrthoMediTec (Industry)
Responsible Party: Dr. Hanna Levy, Clinical Study Consultant, OrthoMediTec
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WF-01
Record Dates: First submitted 2007-08-26; First posted 2007-08-28 (Estimated); Last update posted 2009-01-12 (Estimated); Status verified 2008-02

CONDITIONS: Hip Fracture
Keywords: Hip Prosthesis Implantation
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental)
  Interventions: Device: Intracapsular Femoral Fracture Fixation; Device: WaisFix100i for Intracapsular Femoral Fracture Fixation

INTERVENTIONS:
Device: Intracapsular Femoral Fracture Fixation — The WaisFix100i combines a new and unique Internal Triangular Cage nail fixator and three lag screws.
  Other Names: WaisFix100i
Device: WaisFix100i for Intracapsular Femoral Fracture Fixation — The WaisFix100i combines a new and unique Internal Triangular Cage nail fixator and three lag screws.

SUMMARY:
The purpose of this study is to determine the safety and efficacy of using WaisFix100i device for Intracapsular Femoral Fracture Fixation.

DETAILED DESCRIPTION:
Fractures of the neck of the femur represent an estimated cost to society that exceeds ten billion dollars annually in the USA only.

Fractures have been treated with immobilization, traction, amputation, and internal fixation throughout history. Immobilization by casting, bracing, or splinting a joint above and below the fracture was used for most long bone fractures.

Several studies have suggested that reduction and fixation of an Intracapsular fracture of the hip with multiple pins or screws is associated with a lower rate of morbidity and mortality than treatment with prosthetic replacement. With improved methods of fixation and a tendency toward earlier weight-bearing, internal fixation is believed to be a better mode of treatment for younger, more active patients.

On the other hand, the internal fixation procedure may result with number of possibilities for serious complications and biomechanical disadvantages, leading to the device failure. This led to a growing tendency to prefer total or partial hip replacement as the common treatment for intracapsular fracture, although the internal fixation is the favorable procedure in the professional literature.

OrthoMediTec has developed the WaisFix100i device, a new concept for Intracapsular Femoral Fracture Fixation and bone grafting using minimally invasive procedures. The WaisFix100i combines a new and unique Internal Triangular Cage nail fixator and three lag screws.

The Internal Triangular Cage is inserted into the femoral neck as a strong, solid beam structure to guide and hold the screws in place. The cage supplies the structure to hold the bone graft and screws at the fracture site.

The objectives of this single arm, multi-center, prospective study, are to evaluate the safety and efficacy of using the WaisFix100i device in intracapsular femoral fracture fixation surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Male/Female with Intracapsular femoral fracture type Garden I-II and several III.
2. Age 50 to 75.
3. Subject able to comprehend and give informed consent for participation in this study.

Exclusion Criteria:

1. Known active infectious disease.
2. Terminal diseases
3. Patients in high risk and/or acute cardio-vascular disease.
4. Known cognitive disorder, psychiatric and/or neurological disease
5. Physician objection.
6. Age under 50 or above 75.
7. Concurrent participation in any other clinical study
8. Patients cannot understand or not willing to sign the informed consent.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-09; Primary Completion 2008-03 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
The safety endpoint is measure by paucity incidence of treatment related major complications. | Study duration

SECONDARY OUTCOMES:
Efficacy endpoint is measure by the following: 1. A subject is scored a success if he had no revision surgery, hemi- arthroplasty or total hip replacement surgery by 12 months; 2. Time to functional recovery | Study duration

CONTACTS AND LOCATIONS:
Overall Officials: Marc Waisman, Dr., Principal Investigator — Carmel medical Center, Haifa Israel
Locations (1):
- carmel Medical Center, Haifa, Israel